CLINICAL TRIAL: NCT06003075
Title: Phase II Study of Induction Platinum Doublet in Combination With Nivolumab Followed by Surgery or Concurrent Chemoradiation in Unresectable Stage IIIA-C Non-small Cell Lung Cancer (NSCLC)
Brief Title: Induction Chemo-Nivo in Unresectable Stage III NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Ralph G Zinner (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Ralph G Zinner, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 85869
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer, Nonsmall Cell; Lung Cancer Stage III
Keywords: Nivolumab; unresectable
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Nivolumab; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Chemo, biopsy, surgery with option for post op chemo or no surgery with concurrent chemo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Combination Chemotherapy and Nivolumab and Surgery (Experimental): Patients with lung cancer receiving combination therapy with surgery
  Interventions: Combination Product: Nivolumab and Chemotherapy; Drug: Nivolumab; Procedure: Post Induction Surgery; Radiation: Post Induction XRT
- Combination Chemotherapy and Nivolumab and Radiation (Experimental): Patients with lung cancer receiving combination therapy with radiation
  Interventions: Combination Product: Nivolumab and Chemotherapy; Drug: Nivolumab; Radiation: Post Induction XRT

INTERVENTIONS:
Combination Product: Nivolumab and Chemotherapy — 3 cycles of the proposed nivolumab + platinum doublet (either pemetrexed + carbo/cis or paclitaxel + carbo or docetaxel + carbo/cis for non squamous; or gemcitabine + carbo/cis or paclitaxel + carbo or docetaxel + carbo/cis for squamous) will be administered then CT and biopsy, followed by surgery with option for post-op NIVO-XRT, then 12 cycles NIVO at 480 mg IV every 4 weeks for 12 weeks
Drug: Nivolumab — Participants will receive NIVO at 480 mg IV every 4 weeks for 12 cycles after either surgery or treated with concurrent chemotherapy-nivolumab-radiation
  Other Names: NIVO
Procedure: Post Induction Surgery — Induction Chemo-NIVO x 3 cycles then CT and biopsy, followed by surgery in patients whose tumors were unresectable stage IIIA-C at baseline on the basis of lymphadenopathy and are determined to be resectable after responding to induction chemotherapy-nivolumab. The participants have an option for post op XRT, then will receive NIVO at 480 mg IV every 4 weeks for 12 cycles
  Arms: Combination Chemotherapy and Nivolumab and Surgery
Radiation: Post Induction XRT — Induction Chemo-NIVO x 3 cycles then CT and biopsy, followed by concurrent Chemo and Nivo XRT (60Gy). Participants will receive concurrent thoracic radiation therapy using a standardized 3DCRT or IMRT technique on a linear accelerator operating at 2:6 MV beam energy. The target total dose of thoracic radiation therapy will be 60 Gy in 30 daily fractions of 2 Gy prescribed to the PTV. The participants then will receive NIVO at 480 mg IV every 4 weeks for 12 cycles.

SUMMARY:
The purpose of this study is to determine the response rate, safety, and effectiveness of a combination therapy in patients with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Squamous and non-squamous non-small cell lung cancer that is at baseline, unresectable stage IIIA-IIIC (8th edition AJCC) and not previously treated
* PD-L1 level needs to be measured with values 0-100% eligible
* EGFR/ALK/ROS1 Wild Type or unknown genetic alterations in these genes
* ECOG Performance Status ≤ 1
* Adequate organ and marrow function
* Adequate pulmonary reserve (e.g., FVC, FEV1, TLC, FRC, and DLCO) capable of tolerating the proposed lung resection
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Clinical risk assessment of cardiac function using the New York Heart Association Functional Classification class 2B or better
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have participated in a study with an investigational agent or device within 2 weeks of enrollment
* Any prior radiotherapy to the lung
* Any prior treatment for NSCLC
* Any prior therapy with anti-PD-1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Any history of a severe hypersensitivity reaction to any monoclonal antibody
* Any history of allergy to the study drug components
* primary tumors involving the esophagus
* pancoast tumors
* Patients cannot have primary tumors which would remain unresectable
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Nivolumab or other agents used in study
* Any active or history of autoimmune disease (including any history of inflammatory bowel disease), or history of syndrome that required systemic steroids or immunosuppressive medications
* Ongoing requirement for systemic corticosteroids greater than the equivalent of prednisone 10mg
* previous malignancies
* history of interstitial lung disease
* Patients requiring continuous supplemental oxygen
* Use of any live vaccines against infectious diseases (e.g., influenza, varicella. etc.) within 4 weeks (28 days) of initiation of study therapy
* Active systemic infection requiring therapy
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Zinner, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Groups:
- Combination Chemotherapy and Nivolumab and Surgery: Patients with lung cancer receiving combination therapy with surgery
  Nivolumab and Chemotherapy: 3 cycles of proposed nivolumab + platinum doublet (either pemetrexed + carbo/cis or paclitaxel + carbo or docetaxel + carbo/cis for non squamous; or gemcitabine + carbo/cis or paclitaxel + carbo or docetaxel + carbo/cis for squamous) administered then CT + biopsy, followed by surgery with option for post-op NIVO-XRT, then 12 cycles NIVO at 480 mg IV every 4 weeks for 12 weeks
  Nivolumab: Participants receive NIVO at 480 mg IV every 4 weeks for 12 cycles after either surgery or treated with concurrent chemotherapy-nivolumab-radiation
  Post Induction Surgery: Induction Chemo-NIVO x 3 cycles then CT + biopsy, followed by surgery in patients with unresectable stage IIIA-C tumors at baseline on the basis of lymphadenopathy and determined to be resectable after responding to induction chemotherapy-nivolumab. participants have an option for post op XRT, then NIVO at 480 mg IV every 4 weeks for 12 cycles
  Post Induction XRT: Induction Chemo-NIVO x 3 cycles then CT and biopsy, followed by concurrent Chemo and Nivo XRT (60Gy). Participants will receive concurrent thoracic radiation therapy using a standardized 3DCRT or IMRT technique on a linear accelerator operating at 2:6 MV beam energy. The target total dose of thoracic radiation therapy will be 60 Gy in 30 daily fractions of 2 Gy prescribed to the PTV. Participants then receive NIVO at 480 mg IV every 4 weeks for 12 cycles.
Period: Overall Study
Arm/Group | Combination Chemotherapy and Nivolumab and Surgery | Combination Chemotherapy and Nivolumab and Radiation
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: he study was terminated. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Chemotherapy and Nivolumab and Surgery | Combination Chemotherapy and Nivolumab and Radiation | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Response Rate After Induction
Description: post induction radiographic response by cat scan
Time Frame: 9 weeks
Population: as for baseline characteristics
Arm/Group | Combination Chemotherapy and Nivolumab and Surgery | Combination Chemotherapy and Nivolumab and Radiation
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Toxicity
Description: To assess safety, investigators will evaluate the rate of toxicity as defined by the Common Toxicity Criteria for Adverse Effects (CTCAE) scoring system.
Time Frame: through study completion, up to 18 months
Population: The study was terminated. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Combination Chemotherapy and Nivolumab and Surgery | Combination Chemotherapy and Nivolumab and Radiation
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percent of Participants Receiving Surgery
Description: Rate of converting non-surgical stage III(A-C) to surgically resectable disease
Time Frame: date of surgery, approximately 10 weeks
Population: as for outcome 2
Arm/Group | Combination Chemotherapy and Nivolumab and Surgery | Combination Chemotherapy and Nivolumab and Radiation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pathologic Complete Response (pCR)
Description: Number of participants with Pathologic Complete Response. Pathologic complete response (pCR) is defined by a surgical pathology specimen
Time Frame: post surgery, approximately 10 weeks
Population: as for outcome 2
Arm/Group | Combination Chemotherapy and Nivolumab and Surgery | Combination Chemotherapy and Nivolumab and Radiation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Major Pathological Response (MPR)
Description: MPR rate, defined as number of participants with ≤ 10% residual tumor in lung and lymph nodes
Time Frame: post surgery, approximately 10 weeks
Population: as for outcome 2
Arm/Group | Combination Chemotherapy and Nivolumab and Surgery | Combination Chemotherapy and Nivolumab and Radiation
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of disease progression or death, whichever occurs first.
Time Frame: 2 years
Population: as for outcome 2
Arm/Group | Combination Chemotherapy and Nivolumab and Surgery | Combination Chemotherapy and Nivolumab and Radiation
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Overall Survival (OS)
Description: defined as the duration of time from start of treatment to time of death
Time Frame: 2 years
Population: as for outcome 2
Arm/Group | Combination Chemotherapy and Nivolumab and Surgery | Combination Chemotherapy and Nivolumab and Radiation
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Patient-reported Quality of Life as Measured by FACT-TOI
Description: patient-reported Quality of Life as measured by FACT-TOI (Functional Assessment of Cancer Therapy - Trial Outcome Index); defined as the sum of the scores of the Physical Well-Being (PWB), Functional Well-Being (FWB), and LCS. PWB, FWB, and LCS (lung cancer scale) scores obtained from 7-item questionnaires from the FACT-L (Version 4.0). Questions are on a 5-point scale from 0-4, where 0 = "not at all" and 4 = "very much." Scores range from 0 to 84; higher score indicates better physical aspects of quality of life (QoL).
Time Frame: through study completion, up to 18 months
Population: as for outcome 2
Arm/Group | Combination Chemotherapy and Nivolumab and Surgery | Combination Chemotherapy and Nivolumab and Radiation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The study was terminated. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Description: The study was terminated. Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Combination Chemotherapy and Nivolumab and Surgery | Combination Chemotherapy and Nivolumab and Radiation
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT06003075/Prot_SAP_000.pdf